CLINICAL TRIAL: NCT06291207
Title: A Randomization, Double-blind, Active-controlled, Multicenter, Phase 3 Trial to Evaluate the Efficacy and Safety of AD-224A and AD-224B in Patients with Essential Hypertension
Brief Title: A Study to Evaluate the Efficacy and Safety of AD-224
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-224P3
Record Dates: First submitted 2024-02-27; First posted 2024-03-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AD-224A (Experimental): AD-224A+Placebo of AD-224B+Placebo of AD-224C
  Interventions: Drug: AD-224A; Drug: Placebo of AD-224B; Drug: Placebo of AD-224C
- AD-224B (Experimental): Placebo of AD-224A+AD-224B+Placebo of AD-224C
  Interventions: Drug: AD-224B; Drug: Placebo of AD-224A; Drug: Placebo of AD-224C
- AD-224C (Active Comparator): Placebo of AD-224A+Placebo of AD-224B+AD-224C
  Interventions: Drug: AD-224C; Drug: Placebo of AD-224A; Drug: Placebo of AD-224B

INTERVENTIONS:
Drug: AD-224A — PO, Once daily, 8weeks
  Arms: AD-224A
Drug: AD-224B — PO, Once daily, 8weeks
  Arms: AD-224B
Drug: AD-224C — PO, Once daily, 8weeks
  Arms: AD-224C
Drug: Placebo of AD-224A — PO, Once daily, 8weeks
  Arms: AD-224B; AD-224C
Drug: Placebo of AD-224B — PO, Once daily, 8weeks
  Arms: AD-224A; AD-224C
Drug: Placebo of AD-224C — PO, Once daily, 8weeks
  Arms: AD-224A; AD-224B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AD-224

DETAILED DESCRIPTION:
Condition or disease : Essential Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients with Essential Hypertension
* Other inclusions applied

Exclusion Criteria:

* Patient with Secondary Hypertension
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change rate of MSSBP | Baseline, Week 8
  Change from baseline in mean sitting systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: InHo Chae, M.D., Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No